CLINICAL TRIAL: NCT05214885
Title: Novel Biomarkers of Hypoxia and Metabolism in Clear Cell Renal Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, associate professor, Qianfoshan Hospital
Other Study IDs: CT2021-11-23
Record Dates: First submitted 2022-01-05; First posted 2022-01-31 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: clear cell renal cell carcinoma; carbonic anhydrase IX; HILPDA; NDUFA4L2; ANGPTL4; Cell-free DNA methylomes; EGLN3
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and tumor tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- the ccRCC patient group: The age and gender of patients are not limited. The patient was preliminarily diagnosed as renal carcinoma by imaging examination and finally diagnosed as clear cell renal cell carcinoma by pathology.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study
- the healthy control group: The age and sex of the healthy control group were matched with that of ccRCC patient group. There was no tumor in the kidney or other parts of the body, and no tumor in the blood system. The healthy control group did not have any renal benign diseases, such as kidney stones, diabetic nephropathy, inflammation, and uremia. There are no inflammatory diseases in other parts of the body. The functions of the liver, kidney, and heart were normal.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study
- the benign kidney disease group: The age and sex of this group were matched with that of ccRCC patient group. The patient did not have any tumor but had one of the benign kidney diseases, such as kidney stones, diabetic nephropathy, inflammation, and uremia. The functions of the liver and heart were normal.
  Interventions: Diagnostic Test: No intervention was required for patients or control group in this study

INTERVENTIONS:
Diagnostic Test: No intervention was required for patients or control group in this study — The patient was treated normally and no intervention was required in this study

SUMMARY:
Renal cell carcinoma (RCC) is one of the common malignant tumors in human beings and originates from the renal tubular epithelium. Clear cell renal cell carcinoma (ccRCC) is the main pathological type of RCC. Due to the lack of reliable biomarkers and clinical symptoms for early diagnosis, imaging findings such as ultrasound and CT are needed. When the patients presented typical symptoms, for example, hematuria, backache, and abdominal mass, some of them are in advanced stages of cancer. About a quarter of patients had metastasis at the first diagnosis, and the 5-year survival rate of these patients was less than 10%. Therefore, the early diagnosis of ccRCC and the prevention of tumor recurrence and metastasis are of great significance.

The preliminary studies suggested that some hypoxia and metabolism-related molecules were highly expressed in ccRCC tumors but low in normal kidney tissues. The molecules included carbonic anhydrase IX/9 (CA IX/CA9), the mitochondrial NADH dehydrogenase [ubiquinone] 1 alpha subcomplex, 4-like 2(NDUFA4L2), angiopoietin-like protein 4(ANGPTL4), hypoxia inducible lipid droplet-associated (HILPDA）, and egl-9 family hypoxia-inducible factor 3( EGLN3) et al . Cell-free DNA methylomes were also highly expressed in the blood of ccRCC patients.

In order to further verify the expression status of the above novel biomarkers in ccRCC, the investigators will detect the expressions of these molecules in the tumor and adjacent tissues from 140 ccRCC patients by RT-PCR, Western blot, and immunohistochemistry.140 healthy people were selected as the control group. 30 patients with benign kidney diseases were selected as another control group. Blood and urine samples from the ccRCC group and the control group were collected. The mRNA and protein levels of the above molecules in blood or urine samples were detected by qRT-PCR and ELISA. The correlation between the expression of the above new biomarkers and clinical data, such as early diagnosis, pathological grade, recurrence and metastasis, and survival time, was statistically analyzed. The above molecular changes were dynamically detected before surgery, 1 week, and 6 months after surgery. A receiver-operating characteristic curve (ROC) was used to determine the threshold value of these biomarkers for the diagnosis of renal clear cell carcinoma.

The study is to explore the specific tumor biomarker spectrum for clinical diagnosis, evaluation of recurrence, metastasis, and prognosis of ccRCC, which will be auxiliary early screening and diagnosis, reducing the harm of renal cancer to human health.

ELIGIBILITY:
Inclusion Criteria:

* The age and sex of the healthy control group were matched with that of ccRCC patient group. There was no tumor in the kidney or other parts of the body, and no tumor in the blood system. The healthy control group did not have any renal benign diseases, such as kidney stones, diabetic nephropathy, inflammation, and uremia. There are no inflammatory diseases in other parts of the body; the functions of the liver, kidney, and heart were normal.

Exclusion Criteria:

* The volunteer has tumors in the kidney or other parts of the body, or blood system tumors; The volunteer has benign kidney diseases, such as kidney stones, diabetic nephropathy, nephritis and uremia, etc; The patient has inflammatory disease elsewhere. If the volunteer has any one of the above diseases, it shall be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient was preliminarily diagnosed as renal carcinoma by imaging examination and finally diagnosed as clear cell renal cell carcinoma by pathology. The patient was treated normally and no intervention was required in this study.
  There is no need to collect additional samples. A small part of the remaining samples from routine biochemical and pathological tests of patients can be enough to complete the detections required by the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of novel biomarkers in ccRCC patients before surgery | For ccRCC patients, these six novel biomarkers were detected 1 to 3 days before surgery
  1. The expressions of novel biomarkers in blood samples: The protein levels of CA9, NDUFA4L2, ANGPTL4, HILPDA and EGLN3 in blood samples were detected by ELISA method. The levels of cell-free DNA methylomes in blood samples were detected by real-time fluorescence quantitative PCR method.
  2. The expressions of novel biomarkers in urine samples: The levels of cell-free DNA methylomes in urine samples were detected by real-time fluorescence quantitative PCR method.
Detection of novel biomarkers in ccRCC patients 1 week after surgery | For ccRCC patients, the detection of these biomarkers were completed within one week after surgery
  1. The expressions of novel biomarkers in tissues: In the tumor and adjacent tissues from ccRCC patients, the mRNA expressions of CA9, NDUFA4L2, ANGPTL4, HILPDA and EGLN3 were measured by real-time fluorescence quantitative PCR method. The protein expressions of these five molecules were detected by western blot, and immunohistochemistry methods.
  2. The expressions of novel biomarkers in blood samples: The protein levels of CA9, NDUFA4L2, ANGPTL4, HILPDA and EGLN3 in blood samples were detected by ELISA method. The levels of cell-free DNA methylomes in blood samples were detected by real-time fluorescence quantitative PCR method.
  3. The expressions of novel biomarkers in urine samples: The levels of cell-free DNA methylomes in urine samples were detected by real-time fluorescence quantitative PCR method.
Detection of novel biomarkers in ccRCC patients at 6 months after surgery | For ccRCC patients, these six novel biomarkers were detected at 6 months postoperatively
  1. The expressions of novel biomarkers in blood samples: The protein levels of CA9, NDUFA4L2, ANGPTL4, HILPDA and EGLN3 in blood samples were detected by ELISA method. The levels of cell-free DNA methylomes in blood samples were detected by real-time fluorescence quantitative PCR method.
  2. The expressions of novel biomarkers in urine samples: The levels of cell-free DNA methylomes in urine samples were detected by real-time fluorescence quantitative PCR method.
Detection of novel biomarkers in the control groups as baseline | For the healthy control group and the benign kidney disease group, the levels of these six biomarkers were detected as baseline.
  1. The expressions of novel biomarkers in blood samples: The protein levels of CA9, NDUFA4L2, ANGPTL4, HILPDA and EGLN3 in blood samples were detected by ELISA method. The levels of cell-free DNA methylomes in blood samples were detected by real-time fluorescence quantitative PCR method.
  2. The expressions of novel biomarkers in urine samples: The levels of cell-free DNA methylomes in urine samples were detected by real-time fluorescence quantitative PCR method.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Dr., Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) until the project is completed. Sharing IPD may be available 1 year after publication.

REFERENCES:
- [Background] Moch H, Cubilla AL, Humphrey PA, Reuter VE, Ulbright TM. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part A: Renal, Penile, and Testicular Tumours. Eur Urol. 2016 Jul;70(1):93-105. doi: 10.1016/j.eururo.2016.02.029. Epub 2016 Feb 28. PMID 26935559
- [Background] Rini BI, Campbell SC, Escudier B. Renal cell carcinoma. Lancet. 2009 Mar 28;373(9669):1119-32. doi: 10.1016/S0140-6736(09)60229-4. Epub 2009 Mar 5. PMID 19269025
- [Background] Lucarini L, Magnelli L, Schiavone N, Crisci A, Innocenti A, Puccetti L, Cianchi F, Peri S, Supuran CT, Papucci L, Masini E. Plasmatic carbonic anhydrase IX as a diagnostic marker for clear cell renal cell carcinoma. J Enzyme Inhib Med Chem. 2018 Dec;33(1):234-240. doi: 10.1080/14756366.2017.1411350. PMID 29251173
- [Background] Tello D, Balsa E, Acosta-Iborra B, Fuertes-Yebra E, Elorza A, Ordonez A, Corral-Escariz M, Soro I, Lopez-Bernardo E, Perales-Clemente E, Martinez-Ruiz A, Enriquez JA, Aragones J, Cadenas S, Landazuri MO. Induction of the mitochondrial NDUFA4L2 protein by HIF-1alpha decreases oxygen consumption by inhibiting Complex I activity. Cell Metab. 2011 Dec 7;14(6):768-79. doi: 10.1016/j.cmet.2011.10.008. Epub 2011 Nov 17. PMID 22100406
- [Background] Papandreou I, Cairns RA, Fontana L, Lim AL, Denko NC. HIF-1 mediates adaptation to hypoxia by actively downregulating mitochondrial oxygen consumption. Cell Metab. 2006 Mar;3(3):187-97. doi: 10.1016/j.cmet.2006.01.012. PMID 16517406
- [Background] Liu L, Lan G, Peng L, Xie X, Peng F, Yu S, Wang Y, Tang X. NDUFA4L2 expression predicts poor prognosis in clear cell renal cell carcinoma patients. Ren Fail. 2016 Sep;38(8):1199-205. doi: 10.1080/0886022X.2016.1208517. Epub 2016 Jul 25. PMID 27453328
- [Background] Miikkulainen P, Hogel H, Seyednasrollah F, Rantanen K, Elo LL, Jaakkola PM. Hypoxia-inducible factor (HIF)-prolyl hydroxylase 3 (PHD3) maintains high HIF2A mRNA levels in clear cell renal cell carcinoma. J Biol Chem. 2019 Mar 8;294(10):3760-3771. doi: 10.1074/jbc.RA118.004902. Epub 2019 Jan 7. PMID 30617181
- [Background] Povero D, Johnson SM, Liu J. Hypoxia, hypoxia-inducible gene 2 (HIG2)/HILPDA, and intracellular lipolysis in cancer. Cancer Lett. 2020 Nov 28;493:71-79. doi: 10.1016/j.canlet.2020.06.013. Epub 2020 Aug 18. PMID 32818550
- [Background] Galaup A, Cazes A, Le Jan S, Philippe J, Connault E, Le Coz E, Mekid H, Mir LM, Opolon P, Corvol P, Monnot C, Germain S. Angiopoietin-like 4 prevents metastasis through inhibition of vascular permeability and tumor cell motility and invasiveness. Proc Natl Acad Sci U S A. 2006 Dec 5;103(49):18721-6. doi: 10.1073/pnas.0609025103. Epub 2006 Nov 27. PMID 17130448
- [Background] Nuzzo PV, Berchuck JE, Korthauer K, Spisak S, Nassar AH, Abou Alaiwi S, Chakravarthy A, Shen SY, Bakouny Z, Boccardo F, Steinharter J, Bouchard G, Curran CR, Pan W, Baca SC, Seo JH, Lee GM, Michaelson MD, Chang SL, Waikar SS, Sonpavde G, Irizarry RA, Pomerantz M, De Carvalho DD, Choueiri TK, Freedman ML. Detection of renal cell carcinoma using plasma and urine cell-free DNA methylomes. Nat Med. 2020 Jul;26(7):1041-1043. doi: 10.1038/s41591-020-0933-1. Epub 2020 Jun 22. PMID 32572266